CLINICAL TRIAL: NCT04617886
Title: The Effect of Mood Induction Procedure of Sadness (vs. Joy) in Body Image Through Virtual Reality
Brief Title: The Effect of Mood Induction in Body Image Through Virtual Reality
Acronym: EMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1127840
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-11

CONDITIONS: Sadness; Happiness

STUDY DESIGN:
Intervention Model Description: Within subjects design. Each participant will be tested, in a counterbalanced way, through both (sadness vs. joy) conditions
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sadness condition (Experimental)
  Interventions: Other: Sadness induction; Other: Happiness induction
- Happiness condition (Experimental)
  Interventions: Other: Sadness induction; Other: Happiness induction

INTERVENTIONS:
Other: Sadness induction — Sadness state will be induced with a Virtual Reality program. Mood induction will be done with an emotional induction procedure in virtual reality (Mood induction parks (Baños et al., 2006)). This technique has proven to be effective in previous studies (e.g., van Strien et al. 2013). Virtual reality software simulates an urban park and includes several methods of sadness induction: Velten's tasks (1968) (sentence formulations with negative content about the self; for example, "I am not valuable", "I see no future"); visualization of a image bank with emotional content from the international system of emotional images (IAPS, Lang et al.,1999); listening to a piece of music and viewing a film scene that demonstrated his effectiveness in inducing positive affect (Donen et al. 1952; Eich and Metcalfe 1989; Gross and Levenson 1995), and an autobiographical memory test.
Other: Happiness induction — Happiness state will be induced with a Virtual Reality program. Mood induction will be done with an emotional induction procedure in virtual reality (Mood induction parks (Baños et al., 2006)). This technique has proven to be effective in previous studies (e.g., van Strien et al. 2013). Virtual reality software simulates an urban park and includes several methods of sadness induction: Velten's tasks (1968) (sentence formulations with negative content about the self; for example, "I am not valuable", "I see no future"); visualization of a image bank with emotional content from the international system of emotional images (IAPS, Lang et al.,1999); listening to a piece of music and viewing a film scene that demonstrated his effectiveness in inducing positive affect (Donen et al. 1952; Eich and Metcalfe 1989; Gross and Levenson 1995), and an autobiographical memory test.

SUMMARY:
The effect of emotional induction of sadness (vs. joy) on the mental representation of the body image through the virtual reality

DETAILED DESCRIPTION:
The general objective of this study is to analyze the impact of emotional induction (sadness vs. joy) on the two dimensions (perceptive and affective) of body image with the help of virtual reality. Thus, it is hypothesized that a negative emotional induction may partially explain the change in body image measures.

ELIGIBILITY:
Inclusion Criteria for CLINICAL population:

* ED diagnosis: Anorexia Nervosa, Bulimia Nervosa or Eating Disorder Not Otherwise Specified
* BDI-II - depression symptomatology scores <29 (for ethical reasons)
* Age between 13 and 18

Exclusion Criteria for CLINICAL population:

* suicide risk: the decision of the psychiatrist/psychologist
* present any medical illness or physical incapacity that could impede the experiment
* diagnosis of Binge Eating Disorder
* Body Mass Index <14 or > 28
* pregnancy

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the Body image dissatisfaction state | Baseline; inmediately after procedure
  Body Image States Scale (BISS; Cash, Fleming, Alindogan, Steadman y Whitehead, 2002).
  This is a 6-item self-report questionnaire that measures the individuals' evaluation and affect about their physical appearance (e.g., body image appraisal and satisfaction, as well as emotional experiences) at a particular moment in time: (1) satisfaction with one's overall physical appearance, (2) satisfaction with one's body size and shape, (3) satisfaction with one's weight; (4) feelings of physical attractiveness; (5) current feelings about one's looks relative to how one usually feels; and (6) evaluation of one's appearance relative to how the average person looks. Items are rated on a 9-point bipolar Likert scale. The measure is the composite mean of the items, and higher scores reflect a more favorable body image satisfaction state. The BISS was acceptably internally consistent in the original validation. A Spanish version was translated by the authors of the study.
Change in the Body image estimation | Baseline; inmediately after procedure
  Software Cognitive (developed at the lab) measuring real and ideal body size estimation based on Glendhill et al. (2017) and using Virtual Reality. The results will be reflected as Body Mass Index change (estimation of the own body size and the ideal body size in BMI).
  In the present study, a total of 31 female avatars with different BMI were developed.
  The VR evaluation program allowed for tasks to be performed to estimate the body size (for one's own body and for the ideal body). The body size estimation tasks consisted of two phases. In the first phase, 8 avatars with a different BMI ranging from 14.5 to 28.5 were presented randomly. Ten repetitions were performed for each avatar. In the second phase, 5 avatars were shown with a BMI greater and less in 2 units to the cut-off point estimated in the first phase of the estimation task. Five repetitions were performed for each avatar.

SECONDARY OUTCOMES:
Change in the Positive and negative affect | Baseline; inmediately after procedure
  (PANAS; Watson, Clark, and Tellegen, 1988; Spanish adaptation by López-Gómez, Hervás y Vázquez, 2015).The instrument consists of two scales: positive affection scale (PA) and negative affection scale (NA), each consisting of 10 items. The items are scored using a five-point Likert scale (1 = not at all or very slightly to 5 = very much) in the specified time period (in this study: "right now"). The total score corresponding to the presence of a specific affection, between 10 and 50, is obtained with the sum of the scores of each of the items on the scale. In the Spanish adaptation of the instrument, by López-Gómez, Hervás and Vázquez (2015), the Cronbach alpha coefficient was .92 for the PA and .88 for the AN. While the item-total correlations of the AP factor oscillate between .67 and .74, while those of the AN factor oscillate between .52 and .69.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain